CLINICAL TRIAL: NCT05890794
Title: Open-Label Pilot Trial to Evaluate the Effects of Ilofotase Alfa on Biomarkers in Adult Patients With Hypophosphatasia
Brief Title: Pilot Trial of Single Dose Ilofotase Alfa in Hypophosphatasia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: AM-Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AP-recAP-HPP-01-01
Record Dates: First submitted 2023-05-10; First posted 2023-06-06 (Actual); Results first posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Hypophosphatasia
Keywords: Enzyme replacement therapy
MeSH Terms: conditions — Hypophosphatasia

STUDY DESIGN:
Intervention Model Description: 2 doses will be compared
Masking Description: Trial is masked for received dose; type of drug received is open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 0.8 mg/kg ilofotase alfa (Experimental): Single dose administered intravenously over 1 hour
  Interventions: Biological: Ilofotase Alfa, 0.8 mg/kg
- 3.2 mg/kg ilofotase alfa (Experimental): Single dose administered intravenously over 1 hour
  Interventions: Biological: Ilofotase Alfa, 3.2 mg/kg

INTERVENTIONS:
Biological: Ilofotase Alfa, 0.8 mg/kg — Biological: single 1-hour intravenous infusion of 0.8 mg/kg ilofotase alfa
  Other Names: recAP
  Arms: 0.8 mg/kg ilofotase alfa
Biological: Ilofotase Alfa, 3.2 mg/kg — Biological: single 1-hour intravenous infusion of 3.2 mg/kg ilofotase alfa
  Other Names: recAP
  Arms: 3.2 mg/kg ilofotase alfa

SUMMARY:
The goal of this clinical trial is to compare the effectiveness of two doses of ilofotase alfa, an enzyme replacement treatment, in patients with hypophosphatasia (HPP). The main question it aims to answer is if the harmful accumulating levels of extracellular inorganic pyrophosphate (PPi) and pyridoxal 5'-phosphate (PLP) can be reduced with ilofotase alfa.

Researchers will compare the two doses of ilofotase alfa to see if treatment effects differ between the doses.

DETAILED DESCRIPTION:
Recombinant human alkaline phosphatase (ilofotase alfa) is a full-length human chimeric alkaline phosphatase (ALP) that could benefit patients with hypophosphatasia (HPP), which is characterized by low activity of tissue-nonspecific isoenzyme of alkaline phosphatase (TNSALP).

This is a pilot trial for a potential future trial aimed at identifying whether treatment with ilofotase alfa can normalize circulating levels of PPi, PLP and other biochemical markers of TNSALP deficiency along with the safety/tolerability of different doses of ilofotase alfa. The trial is designed as a single-center, open-label, randomized, parallel group clinical trial in adult patients with HPP. Two different dose levels (0.8 mg/kg and 3.2 mg/kg) of ilofotase alfa will be assessed.

Participants will receive a single dose of ilofotase alfa, administered as a 1-hour intravenous infusion on Study Day 1. Participants will stay at the research center for a total of 12 days; from 2 days before study drug administration (run-in) to 10 days after treatment. An additional follow-up assessment is scheduled 14 days after administration of ilofotase alfa.

Blood and urine samples will be taken daily for drug concentration and laboratory measurements assessing safety and effectiveness of treatment. In addition physical examinations will be performed on Day 1 and as needed afterwards.

ELIGIBILITY:
Inclusion Criteria:

* Genetically confirmed variant in the tissue-nonspecific isozyme alkaline phosphatase (ALPL)-Gene.
* Clinical symptoms of HPP.
* Medical history with 1) at least two independent measures of Alkaline Phosphatase (ALP) below lower level of normal (LLN) and 2) at least one measurement of either PPi or PLP above upper level of normal (ULN).
* Provision of signed and dated informed consent form (ICF) in accordance with local regulations at screening.
* Patients must agree not to get pregnant/not to get their partner pregnant, during the trial. Consequently, patients must agree to use adequate contraception as detailed in study protocol.

Exclusion Criteria:

* Participant is unable or unwilling to participate in all scheduled visits and perform all protocol-mandated assessments.
* Has a known or suspected hypersensitivity to ilofotase alfa or any components of the formulation used.
* Body weight < 40 kilogram and > 120 kilogram.
* Patient has a history of clinically significant abnormalities or of any illness that, in the opinion of the trial investigator, might confound the results of the trial or pose an additional risk to the patient by their participation in the trial.
* NSAID use in the past 2 weeks.
* Use of corticosteroids in the past 4 weeks.
* Use of compounds intended to interfere with bone metabolism (e.g. Denosumab, Teriparatide, Romosozumab, Raloxifene) in the past 3 months.
* Use of bisphosphonates in the past 2 years.
* Participation in a drug trial within 60 days, or five times the half-life of the drug, whichever is longer, prior to administration of ilofotase alfa.
* Use of asfotase alfa in the previous 3 months. Patients will not be withheld from approved asfotase alfa if medically indicated.
* A patient who is currently pregnant or lactating.
* Use of supplements including Vitamin B6.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Seefried, Principal Investigator — Osteologie / Klinische Studieneinheit, Orthopädische Klinik - KLH, Würzburg, Germany
Locations (1):
- Osteologie / Klinische Studieneinheit, Orthopädische Klinik - KLH, Würzburg, Germany

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 12 patients were enrolled, screened and randomized (6 to the 0.8 mg ilofotase alfa dose group, 6 to the 3.2 mg ilofotase alfa dose group)
Groups:
- 0.8 mg/kg Ilofotase Alfa: Single, 1-hour intravenous infusion of 0.8 mg/kg ilofotase alfa
- 3.2 mg/kg Ilofotase Alfa: Single, 1-hour intravenous infusion of 3.2 mg/kg ilofotase alfa
Period: Overall Study
Arm/Group | 0.8 mg/kg Ilofotase Alfa | 3.2 mg/kg Ilofotase Alfa
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intention-to-treat population = all randomized patients
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.8 mg/kg Ilofotase Alfa | 3.2 mg/kg Ilofotase Alfa | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Median (Full Range); unit: years] | 49.5 [41 to 62] | 51.0 [30 to 68] | 51.0 [30 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 3 | 1 | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Maximum Percent Change From Baseline in Extracellular Inorganic Pyrophosphate (PPi)
Description: Percent Change from BaseLine (PCBL) in PPi serum concentration is calculated for all post-dose PPi measures recorded from Day 1 to Day 10. Per patient, 12 measurements were done: 3 at Day 1 and 1 each day from Day 2 to Day 10. The Percent Change from BaseLine for measurement x (x=1,…12) is calculated: PCBL(x)= [(PPi( x)-PPi(baseline))/PPi(baseline)]*100. The subject's maximum percent change from baseline is defined as the Max (PCBL(1), …, PCBL(12)).
Time Frame: Day 1 to Day 10
Population: All randomized patients.
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Overall: Single, 1-hour intravenous infusion of 0.8 mg/kg or 3.2 mg/kg ilofotase alfa
Arm/Group | 0.8 mg/kg Ilofotase Alfa | 3.2 mg/kg Ilofotase Alfa | Overall
Number analyzed (Participants) | 6 | 6 | 12
percent change | -36.46 (11.502) | -77.31 (16.113) | -56.88 (25.165)
Statistical Analysis 1: Comparison: 0.8 mg/kg Ilofotase Alfa vs 3.2 mg/kg Ilofotase Alfa; Analysis of the difference in relative maximum change from baseline between dose groups of ilofotase alfa by a 2-sided t-test for PPi; Test type: Other — The difference in dose group means (0.8 mg/kg - 3.2 mg/kg) was calculated; p = 0.0005, t-test, 2 sided — Significant test: 2-sided; significance level 5%; A 2-sided t-test was carried out to determine whether there is a difference in means between the 0.8 mg/kg and 3.2 mg/kg dose groups; Mean Difference (Final Values) = 40.85, 95% CI 2-sided [22.842 to 58.858]
Statistical Analysis 2: Comparison: 0.8 mg/kg Ilofotase Alfa vs 3.2 mg/kg Ilofotase Alfa; Analysis of the difference in relative maximum change from baseline (LS Means) between dose groups of ilofotase alfa by a mixed model repeated measures (MMRM) analysis for PPi; Test type: Other — The difference between LS Means of change from baseline between dose groups was calculated. The analysis was performed using an MMRM model with fixed effects for baseline value, dose group, timepoint, interaction between dose group and timepoint, as well as random effects for patient and error; p < 0.0001, Mixed Models Analysis — Significant test: 2-sided; significance level 5%; Difference in LS Means = -11.17, 95% CI 2-sided [-16.52 to -5.82], Standard Error of Mean 2.681

2. Primary Outcome: Maximum Percent Change From Baseline in Pyridoxal 5'-Phosphate (PLP)
Description: Percent Change from BaseLine (PCBL) in PLP serum concentration is calculated for all post-dose PLP measures recorded from Day 1 to Day 10. Per patient, 12 measurements were done: 3 at Day 1 and 1 each day from Day 2 to Day 10. The Percent Change from BaseLine for measurement x (x=1,…12) is calculated: PCBL(x)= [(PLP( x)-PLP(baseline))/PLP(baseline)]*100. The subject's maximum percent change from baseline is defined as the Max (PCBL(1), …, PCBL(12)).
Time Frame: Day 1 to Day 10
Population: All randomized patients.
Measure: Mean (Standard Deviation); unit: percent change
Groups:
- Overall: Single, 1-hour intravenous infusion of 0.8 mg/kg ilofotase or 3.2 mg/kg ilofotase alfa
Arm/Group | 0.8 mg/kg Ilofotase Alfa | 3.2 mg/kg Ilofotase Alfa | Overall
Number analyzed (Participants) | 6 | 6 | 12
percent change | -34.68 (8.898) | -65.56 (6.559) | -50.12 (17.768)
Statistical Analysis 1: Comparison: 0.8 mg/kg Ilofotase Alfa vs 3.2 mg/kg Ilofotase Alfa; Analysis of the difference in relative maximum change from baseline between dose groups of ilofotase alfa by a 2-sided t-test for PLP; Test type: Other — The difference in dose group means (0.8 mg/kg - 3.2 mg/kg) was calculated; p < 0.0001, t-test, 2 sided — Significant test: 2-sided; significance level 5%; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 30.89, 95% CI 2-sided [20.831 to 40.941]
Statistical Analysis 2: Comparison: 0.8 mg/kg Ilofotase Alfa vs 3.2 mg/kg Ilofotase Alfa; Analysis of the difference in relative maximum change from baseline (LS Means) between dose groups of ilofotase alfa by an MMRM analysis for PLP; Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.0024, Mixed Models Analysis — Significant test: two-sided; significance level 5%; Difference in LS Means = -22.51, 95% CI 2-sided [-35.81 to -9.20], Standard Error of Mean 6.289

3. Other Pre Specified Outcome: Maximum Percent Change From Baseline in Alkaline Phosphatase (ALP) Activity
Description: Percent Change from BaseLine (PCBL) in ALP Activity is calculated for all post-dose ALP measures recorded from Day 2 to Day 10.
  Per patient, 9 measurements were done: 1 each day from Day 2 to Day 10. The Percent Change from BaseLine for measurement x (x=1,…9) is calculated: PCBL(x)= (ALP(x)-ALP(baseline))/ALP(baseline)*100, [x=1,...,9].
  The subject's maximum percent change from baseline is defined as the Max (PCBL(1), …, PCBL(9))
Time Frame: Day 1 to Day 10
Population: All randomized patients.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | 0.8 mg/kg Ilofotase Alfa | 3.2 mg/kg Ilofotase Alfa | Overall
Number analyzed (Participants) | 6 | 6 | 12
percent change | 2685.57 (1492.991) | 7021.23 (2063.878) | 4853.40 (2841.847)
Statistical Analysis 1: Comparison: 0.8 mg/kg Ilofotase Alfa vs 3.2 mg/kg Ilofotase Alfa; Analysis of the difference in relative maximum change from baseline between dose groups of ilofotase alfa by a 2-sided t-test for ALP activity; Test type: Other — The difference in dose group means (0.8 mg/kg - 3.2 mg/kg) was calculated; p = 0.0019, t-test, 2 sided — Significant test: 2-sided; significance level 5%; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -4335.66, 95% CI 2-sided [-6652.753 to -2018.576]

4. Other Pre Specified Outcome: Maximum Percent Change From Baseline in Urine Phosphoethanolamine (PEA)
Description: Percent Change from BaseLine (PCBL) in PEA concentration is calculated for all post-dose PEA measures recorded from Day 2 to Day 10. Per patient, 9 measurements were done: 1 each day from Day 2 to Day 10. The Percent Change from BaseLine for measurement x (x=1,…9) is calculated: PCBL(x)= [(PEA( x)-PEA(baseline))/PEA(baseline)]*100. The subject's maximum percent change from baseline is defined as the Max (PCBL(1), …, PCBL(9)).
Time Frame: Day 1 to Day 10
Population: All randomized patients.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | 0.8 mg/kg Ilofotase Alfa | 3.2 mg/kg Ilofotase Alfa | Overall
Number analyzed (Participants) | 6 | 6 | 12
percent change | -28.58 (15.161) | -51.82 (19.614) | -40.20 (20.573)
Statistical Analysis 1: Comparison: 0.8 mg/kg Ilofotase Alfa vs 3.2 mg/kg Ilofotase Alfa; Analysis of the difference in relative maximum change from baseline between dose groups of ilofotase alfa by a 2-sided t-test for urine PEA; Test type: Other — The difference in dose group means (0.8 mg/kg - 3.2 mg/kg) was calculated; p = 0.0693, t-test, 2 sided — Significant test: 2-sided; significance level 5%; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 23.25, 95% CI 2-sided [-2.319 to 48.812]
Statistical Analysis 2: Comparison: 0.8 mg/kg Ilofotase Alfa vs 3.2 mg/kg Ilofotase Alfa; Analysis of the difference in relative maximum change from baseline (LS Means) between dose groups of ilofotase alfa by an MMRM analysis for urine PEA; Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.7086, Mixed Models Analysis — Significant test: 2-sided; significance level 5%; Difference in LS Means = -8.76, 95% CI 2-sided [-57.88 to 40.35], Standard Error of Mean 22.986

5. Other Pre Specified Outcome: Maximum Percent Change From Baseline in Pyridoxal (PL).
Description: Percent Change from BaseLine (PCBL) in PL serum concentration is calculated for all post-dose PL measures recorded from Day 1 to Day 10. Per patient, 12 measurements were done: 3 at Day 1 and 1 each day from Day 2 to Day 10. The Percent Change from BaseLine for measurement x (x=1,…12) is calculated: PCBL(x)= [(PL( x)-PL(baseline))/PL(baseline)]*100. The subject's maximum percent change from baseline is defined as the Max (PCBL(1), …, PCBL(12)).
Time Frame: Day 1 to Day 10
Population: All randomized patients.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | 0.8 mg/kg Ilofotase Alfa | 3.2 mg/kg Ilofotase Alfa | Overall
Number analyzed (Participants) | 6 | 6 | 12
percent change | 409.76 (138.504) | 222.33 (91.332) | 316.05 (148.635)
Statistical Analysis 1: Comparison: 0.8 mg/kg Ilofotase Alfa vs 3.2 mg/kg Ilofotase Alfa; Analysis of the difference in relative maximum change from baseline between dose groups of ilofotase alfa by a 2-sided t-test for PL; Test type: Other — The difference in dose group means (0.8 mg/kg - 3.2 mg/kg) was calculated; p = 0.0199, t-test, 2 sided — Significant test: 2-sided; significance level 5%; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 187.43, 95% CI 2-sided [36.516 to 338.344]
Statistical Analysis 2: Comparison: 0.8 mg/kg Ilofotase Alfa vs 3.2 mg/kg Ilofotase Alfa; Analysis of the difference in relative maximum change from baseline (LS Means) between dose groups of ilofotase alfa by an MMRM analysis for PL; Test type: Other — [test comment as in outcome 1, analysis 2]; p = 0.2034, Mixed Models Analysis — Significant test: 2-sided; significance level 5%; Difference in LS Means = -12.51, 95% CI 2-sided [-31.92 to 6.89], Standard Error of Mean 9.767

6. Other Pre Specified Outcome: Maximum Fold Change From Baseline in PL/PLP Ratio
Description: Fold Change from BaseLine (FCBL) in PL/PLP ratio is calculated for all post-dose PL/PLP ratio measures recorded from Day 1 to Day 10. Per patient, 12 measurements were done: 3 at Day 1 and 1 each day from Day 2 to Day 10. The Fold Change from BaseLine for measurement x (x=1,…12) is calculated: FCBL(x)= (PL/PLPratio( x) / PL/PLPratio(baseline)). The subject's maximum fold change from baseline is defined as the Max (FCBL(1), …, FCBL(12)).
Time Frame: Day 1 to Day 10
Population: All randomized patients.
Measure: Mean (Standard Deviation); unit: fold change
Arm/Group | 0.8 mg/kg Ilofotase Alfa | 3.2 mg/kg Ilofotase Alfa | Overall
Number analyzed (Participants) | 6 | 6 | 12
fold change | 6.9145 (1.83957) | 7.8062 (2.70554) | 7.3604 (2.25440)
Statistical Analysis 1: Comparison: 0.8 mg/kg Ilofotase Alfa vs 3.2 mg/kg Ilofotase Alfa; Analysis of the difference in fold change from baseline between dose groups of ilofotase alfa by a 2-sided t-test for PL/PLP ratio; Test type: Other — The difference in dose group means (0.8 mg/kg - 3.2 mg/kg) was calculated; p = 0.5195, t-test, 2 sided — Significant test: 2-sided; significance level 5%; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.89, 95% CI 2-sided [-3.868 to 2.084]
Statistical Analysis 2: Comparison: 0.8 mg/kg Ilofotase Alfa vs 3.2 mg/kg Ilofotase Alfa; Analysis of the difference in fold change form baseline (LS Means) between dose levels of ilofotase alfa by an MMRM analysis for PL/PLP ratio; Test type: Other — The difference between LS Means of fold change from baseline between dose groups was calculated. The analysis was performed using an MMRM model with fixed effects for baseline value, dose group, timepoint, interaction between dose group and timepoint, as well as random effects for patient and error; p < 0.0001, Mixed Models Analysis — Significant test: 2-sided; significance level 5%; Difference in LS Means = 1.01, 95% CI 2-sided [0.69 to 1.33], Standard Error of Mean 0.161

7. Other Pre Specified Outcome: Treatment-emergent Adverse Events (TEAEs)
Description: Any untoward medical occurrence in a patient enrolled and treated in the clinical trial regardless of its causal relationship to the trial medication.
Time Frame: Day 1 to Day 15
Population: All patients who received trial medication were included in the population for the safety analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | 0.8 mg/kg Ilofotase Alfa | 3.2 mg/kg Ilofotase Alfa | Overall
Number analyzed (Participants) | 6 | 6 | 12
Participants | 1 | 3 | 4

ADVERSE EVENTS:
Time Frame: Day 1 to Day 15
Groups:
- Overall: Single dose administered intravenously over 1 hour
  Ilofotase Alfa, 0.8 or 3.2 mg/kg: Biological: single 1-hour intravenous infusion of 0.8 or 3.2 mg/kg ilofotase alfa
Arm/Group | 0.8 mg/kg Ilofotase Alfa | 3.2 mg/kg Ilofotase Alfa | Overall
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/12
Other Adverse Events (participants affected / at risk) | 1/6 | 3/6 | 4/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.8 mg/kg Ilofotase Alfa (N=6) | 3.2 mg/kg Ilofotase Alfa (N=6) | Overall (N=12)
Dysgeusia (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Restless arm syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI may publish the study results but must submit the publication to the sponsor for review at least 60 days prior to publication. The sponsor may request changes/removals of sponsor information. The PI should remove such information if the correct presentation of the results is still ensured. The PI must consider the sponsor's other comments but must not adopt them. If publication could affect the patentability of the invention, the sponsor may request an additional period of up to 120 days.

DOCUMENTS (2):
  • Study Protocol (2023-03-30): https://cdn.clinicaltrials.gov/large-docs/94/NCT05890794/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-05): https://cdn.clinicaltrials.gov/large-docs/94/NCT05890794/SAP_001.pdf